CLINICAL TRIAL: NCT07035483
Title: Changes in Adipose and Muscle Tissue Function and Their Impact on Metabolic Health Following Bariatric Surgery
Brief Title: Changes in Fat and Muscle Tissue Function and Their Impact on Metabolic Health After Bariatric Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Shaihong Zhu (Other)
Responsible Party: Sponsor-Investigator, Shaihong Zhu, Chief of Metabolic and Bariatric Surgery, Xiangya Third Hospital, Central South University, The Third Xiangya Hospital of Central South University
Organization: The Third Xiangya Hospital of Central South University (Other)
Other Study IDs: 2024552
Record Dates: First submitted 2025-06-08; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Obesity-related Medical Conditions; Sarcopenic Obesity; Adipose Tissue, Abdominal
Keywords: Obesity; Ectopic Fat Deposition; Sarcopenic Obesity; Bariatric Surgery; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric surgery — This is a prospective observational study evaluating the metabolic and tissue-level effects of bariatric surgery in obese individuals. The intervention includes either laparoscopic sleeve gastrectomy (LSG) or Roux-en-Y gastric bypass (RYGB), performed according to standard clinical guidelines. No experimental procedures are added beyond routine care. Skeletal muscle quality and visceral fat distribution are assessed using MRI and clinical biomarkers at multiple postoperative time points (baseline, 3 months, 12 months, and annually up to 5 years). A healthy control group undergoes baseline evaluation only, without surgical intervention.

SUMMARY:
This prospective, single-center observational cohort study aims to explore the relationship between skeletal muscle quality, fat distribution, and metabolic health in Chinese patients with obesity, and to evaluate how bariatric surgery influences these parameters.

A total of 120 participants will be enrolled, including 60 patients undergoing bariatric surgery and 60 age- and sex-matched healthy controls. The study involves cross-sectional comparisons of ectopic fat and muscle composition, as well as longitudinal follow-up of surgical patients at multiple time points up to 5 years postoperatively.

MRI will be used to quantify regional fat and muscle composition, while metabolic parameters, inflammatory markers, and gut microbiota profiles will also be assessed. Primary outcomes include skeletal muscle mass and fat infiltration, visceral and subcutaneous fat volumes, and changes in insulin resistance.

This study seeks to clarify the mechanisms by which bariatric surgery improves metabolic function and to identify early changes in muscle-fat composition that may predict long-term metabolic outcomes.

ELIGIBILITY:
Inclusion Criteria (For Surgical Group):

* Aged 18 to 65 years (inclusive)
* Meets clinical criteria for sleeve gastrectomy or Roux-en-Y gastric bypass surgery
* Willing and able to comply with study procedures and follow-up visits Capable of understanding and signing the informed consent form

Inclusion Criteria (For Healthy Control Group):

* Aged 18 to 65 years (inclusive)
* Body mass index (BMI) between 18.0 and 24.0 kg/m²
* No history of metabolic disorders (e.g., hypertension, type 2 diabetes, fatty liver disease, or dyslipidemia)
* No history of gastrointestinal surgery
* Able to undergo MRI and willing to provide baseline clinical data and biological samples
* Able to understand and sign informed consent

Exclusion Criteria :

* Type 1 diabetes mellitus or latent autoimmune diabetes in adults (LADA)
* History of pancreatitis, gastrointestinal or pancreatic surgery
* Severe complications of type 2 diabetes or major organ dysfunction that may affect surgical safety
* Active alcohol or drug dependence, severe psychiatric illness, cognitive impairment, or suicidal ideation
* Pregnant or breastfeeding women, or women planning pregnancy during the follow-up period
* Contraindications to MRI examination, including:

Cardiac pacemaker Artificial heart valves Ferromagnetic vascular clips Metallic foreign bodies in the eye

∙Considered unsuitable for the study by investigators based on risk-benefit assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult participants aged 18 to 65 years, including two groups: (1) obese patients undergoing bariatric surgery (either sleeve gastrectomy or Roux-en-Y gastric bypass), and (2) healthy individuals with normal BMI (18.0-24.0 kg/m²) and no metabolic comorbidities. The surgical group consists of patients eligible for metabolic surgery based on national clinical guidelines. The healthy control group is matched by age and sex and will undergo only baseline assessments. All participants must be able to provide informed consent and comply with study procedures. The study population is recruited from Xiangya Third Hospital, Central South University.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Skeletal Muscle Fat Infiltration and Quality (measured by MRI) | Baseline, 3 months, 12 months, annually up to 5 years
  Quantitative evaluation of intramuscular fat content using MRI-derived proton density fat fraction (PDFF) and muscle attenuation indices in the thigh and paraspinal muscles. Muscle quality will be assessed by MRI signal intensity and texture features to detect early changes in muscle composition post-surgery.
Change in Visceral and Subcutaneous Fat Volume (measured by MRI) | Baseline, 3 months, 12 months, annually up to 5 years
  MRI-based measurement of visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT), liver fat percentage (LFP), and pancreatic fat percentage (PFP) to track region-specific fat redistribution after bariatric surgery.

SECONDARY OUTCOMES:
Change in fasting glucose | Baseline, 3 months, 12 months, annually up to 5 years
  Fasting glucose to evaluate metabolic improvement after surgery.
Change in HbA1c | Baseline, 3 months, 12 months, annually up to 5 years
  HbA1c to evaluate metabolic improvement after surgery.
Change in triglycerides | Baseline, 3 months, 12 months, annually up to 5 years
  Triglycerides to evaluate metabolic improvement after surgery.
Change in LDL-C | Baseline, 3 months, 12 months, annually up to 5 years
  LDL-C to evaluate metabolic improvement after surgery.
Change in HDL-C | Baseline, 3 months, 12 months, annually up to 5 years
  HDL-C to evaluate metabolic improvement after surgery.
Change in total cholesterol | Baseline, 3 months, 12 months, annually up to 5 years
  total cholesterol to evaluate metabolic improvement after surgery.
Change in insulin resistance | Baseline, 3 months, 12 months, annually up to 5 years
  HOMA-IR to evaluate metabolic improvement after surgery.
Change in body mass index | Baseline, 3 months, 12 months annually up to 5 years
  Body mass index (BMI), calculated as weight in kilograms divided by height in meters squared (kg/m²), will be measured at baseline and follow-up visits to assess changes in overall adiposity after bariatric surgery. BMI will be used as a general anthropometric indicator of weight loss efficacy over time.
Change in waist circumference | Baseline, 3 months, 12 months annually up to 5 years
  Waist circumference will be measured in centimeters using a standardized tape measure at the midpoint between the lowest rib and the iliac crest. This anthropometric indicator will be used to evaluate central (abdominal) fat reduction following bariatric surgery. Measurements will be taken at baseline and at follow-up time points to assess longitudinal changes.
Change in hip circumference | Baseline, 3 months, 12 months annually up to 5 years
  Hip circumference will be measured in centimeters at the widest portion of the buttocks using a standardized measuring tape. This anthropometric measure will help assess changes in fat distribution following bariatric surgery. Measurements will be recorded at baseline and follow-up visits to monitor longitudinal changes in body composition.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Third Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes (e.g., MRI measurements, metabolic indicators, and inflammatory markers) may be shared with qualified researchers upon reasonable request. Data will be made available after publication of the main results and approval by the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication of primary results; available for up to 3 years.
Access Criteria: Requests must be accompanied by a research proposal and data use agreement. Access will be granted to researchers whose proposed use of the data has been approved by the study team.